CLINICAL TRIAL: NCT06892925
Title: QL1706 Combined With Lenvatinib and GEMOX as First - Line Treatment for Unresectable Biliary Tract Tumors: A Single - Arm, Open - Label, Multi - Center, Prospective Phase II Clinical Trial (Spring Study)
Brief Title: QL1706 Combined With Lenvatinib and GEMOX as First - Line Treatment for Unresectable Biliary Tract Tumors
Acronym: Spring
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Feng Zhang, Professor, Eastern Hepatobiliary Surgery Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2025-H011-P001
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Biliary Tract Tumors
Keywords: QL1706; Lenvatinib; GEMOX; First - Line Treatment
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Intervention Model Description: QL1706 combined with lenvatinib and GEMOX
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): QL1706 Combined with Lenvatinib and GEMOX
  Interventions: Drug: QL1706

INTERVENTIONS:
Drug: QL1706 — Eligible participants will receive QL1706 at 5.0 mg/kg intravenously every 3 weeks, lenvatinib at 8 mg orally once daily every 3 weeks, oxaliplatin at 85 mg/m², and gemcitabine at 1000 mg/m² (on days 1 and 8 of each cycle) for up to 8 cycles. Then, they will continue with QL1706 and lenvatinib until clinical progression, imaging progression per RECIST 1.1, unacceptable toxicity, withdrawal of consent, or other discontinuation criteria are met.
  Other Names: Lenvatinib; GEMOX

SUMMARY:
QL1706 Combined with Lenvatinib and GEMOX as First - Line Treatment for Unresectable Biliary Tract Tumors：A Single - Arm, Open - Label, Multi - Center, Prospective Phase II Clinical Trial (Spring Study)

DETAILED DESCRIPTION:
This open - label, prospective, single - arm, multicenter phase II clinical study aims to assess the efficacy and safety of QL1706 combined with lenvatinib and GEMOX as first - line treatment for patients with unresectable biliary tract tumors.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily participates in the trial, provides full informed consent, signs a written consent form, and demonstrates good compliance.
2. The patient is aged 18 or older, regardless of gender.
3. The patient has a histologically confirmed diagnosis of unresectable locally advanced or metastatic biliary tract cancer, including cholangiocarcinoma (intrahepatic and extrahepatic) and gallbladder cancer.
4. The patient is newly diagnosed with unresectable locally advanced or metastatic biliary tract cancer and has not received prior systemic therapy.
5. Patients who have previously received radical treatment (surgery, adjuvant chemotherapy, and/or radiotherapy) are allowed, provided disease recurrence is >6 months after treatment. Those who received adjuvant therapy (chemotherapy and/or radiotherapy) and are >6 months post-treatment are also eligible.
6. At baseline, the patient has at least one measurable lesion according to RECIST v1.1 that can be repeatedly and accurately measured.
7. The patient has an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-1.
8. The patient has an expected survival of ≥12 weeks.
9. The patient has adequate organ and bone marrow function, meeting the following criteria (within 14 days before starting study treatment):

   * Hematology (no transfusions, granulocyte colony-stimulating factor [G-CSF], or corrective medications within 14 days of screening): Hemoglobin (Hb) ≥90 g/L; Absolute Neutrophil Count (ANC) ≥1.5×10⁹/L; Platelets (PLT) ≥75×10⁹/L.
   * Biochemistry (no albumin transfusion within 14 days of screening): Total bilirubin (BIL) ≤2×upper limit of normal (ULN) (≤3×ULN for Gilbert's syndrome patients); Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤3.0×ULN (≤5×ULN for liver metastases patients); Serum creatinine (Cr) ≤1.5×ULN or endogenous creatinine clearance rate ≥50 ml/min (Cockcroft-Gault formula).
   * For males: Cr clearance = ((140 - age) × weight) / (72 × serum Cr)
   * For females: Cr clearance = ((140 - age) × weight) / (72 × serum Cr) × 0.85 (weight in kg; serum Cr in mg/mL).
10. HBV-infected patients (HBsAg and/or anti-HBc positive) with detectable HBV DNA (≥10 IU/mL or above local laboratory detection limit) must receive antiviral therapy before study drug administration, as per institutional practice, to ensure viral suppression. They must continue antiviral therapy during the study and for 6 months after the last dose. Anti-HBc-positive patients without detectable HBV DNA (<10 IU/mL or below detection limit) do not require antiviral therapy unless HBV DNA exceeds 10 IU/mL or the local laboratory detection limit during the study.
11. Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days before the first dose.
12. Women of childbearing potential engaging in sexual activity with non-sterilized males must use acceptable contraception from screening until 120 days after the last study drug dose.
13. Non-sterilized male patients engaging in sexual activity with women of childbearing potential must use effective contraception from screening until 120 days after the last dose. Contraception cessation after this period should be discussed with the investigator.
14. The patient is willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study requirements.

Exclusion Criteria:

1. Cholangiocarcinoma of rare histopathological types confirmed by histology or cytology, such as ampullary cancer, small cell cancer, neuroendocrine tumors, sarcoma, and mucinous cystic tumors.
2. Subjects with other malignancies within 5 years before enrollment, except for basal cell carcinoma of the skin or carcinoma in situ of the cervix that has been cured.
3. History of leptomeningeal carcinoma, brain metastasis.
4. Participation in another interventional clinical study within the past 3 months, or concurrent enrollment in another clinical study, unless it is an observational, non-interventional study or the follow-up period of an interventional study.
5. Any disease evidence deemed by the investigator to disqualify the subject, such as uncontrolled hypertension, active bleeding disorder, active infection, active interstitial lung disease, severe chronic gastrointestinal disease related to diarrhea, psychiatric illness, or social condition, or a history of allogeneic organ transplantation.
6. Severe cardiovascular disease history: NYHA Class II or above heart failure, unstable angina, myocardial infarction, uncontrolled arrhythmia, or cerebrovascular accident within 12 months before drug administration; echocardiogram showing LVEF <50%; QTc >480ms (Fridericia method, average of three consecutive measurements 2 minutes apart if QTc is abnormal); poorly controlled hypertension (systolic BP ≥150 mmHg and/or diastolic BP ≥100 mmHg, based on the average of ≥2 measurements); history of hypertensive crisis or encephalopathy.
7. Active autoimmune disease within the past 2 years or a history of autoimmune disease that may recur, including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, colitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (excluding patients controlled by hormone replacement therapy).
8. Previous immunotherapy, including immune checkpoint inhibitors (e.g., anti-PD-1/L1, CTLA-4, TIGIT, LAG3 antibodies), immune checkpoint agonists (e.g., CD40, CD137, OX40 antibodies), or other immunotherapy for tumor immune mechanisms, except therapeutic antitumor vaccines.
9. Co-infection with HBV (HBsAg and/or anti-HBcAb positive with detectable HBV DNA) and HCV (anti-HCV antibody positive), or HBV and HDV (anti-HDV antibody positive).
10. Severe peptic ulcer, gastritis, gastrointestinal perforation, abdominal fistula, obstruction, intra-abdominal abscess, or acute gastrointestinal hemorrhage within 6 months before first dose; acute exacerbation of COPD within 1 month before first dose.
11. Life-threatening bleeding event within 3 months before first study drug administration, including those requiring transfusion, surgery, local treatment, or ongoing medication.
12. Major surgery or severe trauma within 30 days before first dose, or planned major surgery within 30 days after first dose (investigator's decision); minor local surgery within 3 days before first dose (excluding central venous catheter placement and venous port implantation).
13. Pregnant or breastfeeding women; men or women of reproductive potential unwilling to use effective contraception from screening until 90 days after last study intervention dose or 180 days after last investigational drug dose.
14. Known allergy or hypersensitivity to any study intervention or its excipients.
15. Other patients deemed unsuitable for inclusion by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-06-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 4 years
  ORR was assessed by investigators per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to approximately 4 years
  DCR was assessed by investigators per RECIST 1.1
Time to Response (TTR) | Up to approximately 4 years
  TTR was assessed by investigators per RECIST 1.1
Duration of Response (DOR) | Up to approximately 4 years
  DOR was assessed by investigators per RECIST 1.1
Progression-free Survival (PFS) | Up to approximately 4 years
  PFS was assessed by investigators per RECIST 1.1
12months-PFS rate | 12 months
  12months-PFS rate was assessed by investigators per RECIST 1.1
6months-PFS Rate | 6 months
  6months-PFS Rate was assessed by investigators per RECIST 1.1
Overall Survival (OS) | Up to approximately 4 years
  OS was defined as the time from randomization to death due to any cause.
12months-OS Rate | 12 months
  12months-OS Rate was assessed by investigators per RECIST 1.1
24months-OS Rate | 24 months
  24months-OS Rate was assessed by investigators per RECIST 1.1
Incidence of Adverse Events (AEs) | Up to approximately 4 years
  An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, Principal Investigator — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- the Third Affiliated Hospital of Naval Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No